CLINICAL TRIAL: NCT04654429
Title: Does Higher Operation Theatre Ambient Temperature and Intravenous Ondansetron Prophylaxis Reduce Incidence of Post-spinal Shivering in Obstetric Population? A Double-blind, Randomised, Factorial Study.
Brief Title: Does Higher OT Temperature and IV Ondansetron Reduce Incidence of PSS in Parturients?
Acronym: HOTON
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Lim Siu Min (Other)
Responsible Party: Sponsor-Investigator, Dr Lim Siu Min, Lecturer and Clinical Specialist, University of Malaya
Organization: University of Malaya (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NMRR-20-2158-56283; 202073-8861 (Other: MREC UMMC)
Record Dates: First submitted 2020-11-11; First posted 2020-12-04 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Temperature Change, Body; Chills; Tremor; Nausea, Postoperative; Vomiting, Postoperative; Postoperative Shivering
Keywords: Post-spinal shivering; Subarachnoid block; obstetrics; caesarean section; temperature; ondansetron; factorial study
MeSH Terms: conditions — Body Temperature Changes; Chills; Tremor; Postoperative Nausea and Vomiting | interventions — Ondansetron

STUDY DESIGN:
Intervention Model Description: All patients participating in this study will be randomised two times into 4 groups: LP, HP, LO, HO (L= low-temperature range, H= high-temperature range, P= placebo, O=Ondansetron). The OT temperature will be set to a random range on every Monday, 7am to either lower temperature range group (17.0-19.0⁰C), set at 18.0⁰C; or higher temperature range group (19.1-22.0⁰C), set at 21.0⁰C by an OT engineer who is not involved in this study. OT engineer will open a sealed opaque envelope which contains target temperature to be set for the week, which is randomised prior using computer generated sequence. The temperature setting will maintain for one week and change on the following Monday 7am.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lower OT temperature with placebo (LP) (Placebo Comparator): Lower OT temperature with placebo This group function as a main control arm. Incidence of PSS will be documented usual / standard OT temperature which is 17-19 degree celsius, and without giving any pharmacological intervention to prevent PSS.
  Interventions: Drug: Placebo; Other: Lower OT temperature Range
- Higher OT temperature with placebo (HP) (Active Comparator): Higher OT temperature with placebo This group will receive one non-pharmacological intervention, which is higher OT temperature 19-22 degree celsius. The aim of this intervention is to reduce heat loss therefore incidence of PSS for obstetric population coming for lower segment cesarean section (LSCS) by reducing the temperature gradient between the body and environment.
  Interventions: Other: Higher OT temperature range; Drug: Placebo
- Lower OT temperature with IV Ondansetron 4mg (LO) (Active Comparator): Lower OT temperature with Ondansetron 4mg intravenous. This group also will receive one pharmacological intervention, which is IV ondansetron 4mg to prevent incidence of PSS under standard OT temperature 17-19 degrees.
  Interventions: Drug: IV Ondansetron 4mg; Other: Lower OT temperature Range
- higher OT temperature 19-22 and IV ondansetron 4mg (HO) (Active Comparator): This group will receive 2 interventions - higher OT temperature 19-22 and IV ondansetron 4mg. This group is designed to see if when both intervention combined, will further reduce the incidence of PSS among obstetrics population.
  Interventions: Drug: IV Ondansetron 4mg; Other: Higher OT temperature range

INTERVENTIONS:
Drug: IV Ondansetron 4mg — IV ondansetron 4mg
  Other Names: Pharmacological intervention
  Arms: Lower OT temperature with IV Ondansetron 4mg (LO); higher OT temperature 19-22 and IV ondansetron 4mg (HO)
Other: Higher OT temperature range — OT temperature set to 19-22 degree celsius
  Other Names: Non-pharmacological intervention
  Arms: Higher OT temperature with placebo (HP); higher OT temperature 19-22 and IV ondansetron 4mg (HO)
Drug: Placebo — IV Normal Saline 2cc will be given
  Other Names: Control
  Arms: Higher OT temperature with placebo (HP); Lower OT temperature with placebo (LP)
Other: Lower OT temperature Range — OT temperature set to 17-19 degree celsius
  Other Names: Control
  Arms: Lower OT temperature with IV Ondansetron 4mg (LO); Lower OT temperature with placebo (LP)

SUMMARY:
This study will look at the incidence of post-spinal shivering (PSS) among the obstetrics population and will investigate whether higher operation theater (OT) temperature range or/and IV Ondansetron are able to reduce the incidence of PSS. This is a double-blind, randomized, factorial study, patients will be grouped into 4 groups - LP, HP, LO, HO (L= low-temperature range, H= high-temperature range, P= placebo, O=Ondansetron). All patients undergoing cesarean section under spinal anesthesia will be recruited, and it will be conducted in obstetrics OT.

DETAILED DESCRIPTION:
Many studies have been conducted to look at methods to prevent and treat postspinal shivering. However, there is still no clear protocol or gold standard for post-spinal shivering management. This is due to the fact that post-spinal shivering mechanisms are complex and are broadly grouped into thermoregulatory and non-thermoregulatory. Preventive measures that have been studied are broadly classified into pharmacological methods and non-pharmacological methods. For Non-pharmacological method, active warming of the patient by various methods have been found to be effective in preventing PSS. However, there is no study that looks at ways to reduce heat loss hence maintaining normothermia and preventing PSS in patients. Therefore in this study, we will be investigating if higher OT temperature will reduce the incidence of PSS. As for pharmacological methods, many drugs have been studied for examples analgesics (tramadol), opioid receptor agonists (pethidine, fentanyl), cholinesterase inhibitors (physostigmine), N-methyl-D-aspartate receptor antagonists (ketamine, magnesium sulphate), α2-central agonists (clonidine, dexmedetomidine), antiserotonergic (ondansetron) and anti-inflammatory drugs (dexamethasone). Ondansetron is usually used to prevent chemotherapy or radiotherapy-induced nausea vomiting and Post-operative nausea and vomiting. Due to the fact that it is generally a safe drug and has added benefit as an anti-emetics especially for obstetrics population, this drug is chosen to be studied. We will also look at the efficacy of the combined effect of increased OT temperature and prophylaxis ondansetron on preventing PSS.

ELIGIBILITY:
Inclusion Criteria:

* All elective and emergency obstetric patients who are going for lower segment caesarean section (LSCS) under spinal anaesthesia in UMMC.
* Patient who are given combined spinal epidural anaesthesia (CSE) without epidural local anaesthetic top-up will be included.

Exclusion Criteria:

1. Patients who refused to provide study consent
2. Caesarean section planned under general or epidural anaesthesia or potential conversion to general anaesthesia intraoperatively
3. Royal College of Obstetrics and Gynaecology (RCOG) classification of urgency caesarean section Grade I - Immediate threat to life of woman and child. (29)
4. Patients with psychiatric disorders who are taking selective serotonin reuptake inhibitor (SSRI) and serotonin-noradrenaline reuptake inhibitor (SNRI)
5. Patients who has problems with any types of tremor or involuntary movements and neuromuscular disorders such as Parkinson Disease and muscular dystrophy will be excluded from the study as this will interfere with the clinical interpretation of shivering
6. Patients with history of allergic / hypersensitive reactions towards ondansetron.
7. Patients who received ondansetron intraoperatively as anti-emetics.
8. Recruited patients will be excluded if OT temperature on the day of recruitment does not fulfil the OT temperature range fixed for the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Parturients going for lower segment cesarean section
Enrollment: 628 (Estimated)
Dates: Start 2020-10-13 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
To Demonstrate higher OT temperature range ( 19.1- 22.0 degree Celcius) is effective in reducing the incidence PSS in parturients. | 1 year
  Assessment of patient's shivering grade according to Crossley and Mahajan classification in both Higher temperature range group ( 19.1 -22.0 degree Celcius) compared to lower OT temperature range group (17.0 - 19.0 degree Celcius) Grade 0 - No Shivering Grade 1 - No visible muscle activity, but one or more of piloerection , peripheral vasoconstriction or peripheral cyanosis ( other causes excluded) Grade 2 - Muscular activity in only one muscle group Grade 3 - Moderate muscle activity in more than one muscle group but not generalised shaking Grade 4 - Violent muscular that involves the entire body
To demonstrate IV Ondansetron is effective in reducing the incidence of PSS in parturient undergoing LSCS. | 1 year
  Assessment of patient's shivering grade according to Crossley and Mahajan classification in both patients receiving placebo group vs receiving Ondansetron group:
  Grade 0 - No Shivering Grade 1 - No visible muscle activity, but one or more of piloerection , peripheral vasoconstriction or peripheral cyanosis ( other causes excluded) Grade 2 - Muscular activity in only one muscle group Grade 3 - Moderate muscle activity in more than one muscle group but not generalised shaking Grade 4 - Violent muscular that involves the entire body

SECONDARY OUTCOMES:
To determine the incidence of PSS | 1 year
  Number patients of with shivering grade 3 and above.
To determine the average threshold body temperature, ⁰C at which shivering occur. | 1 year
  To determine the average range of temperature that grade 3 and above shivering occurred among the recruited population from linear graph
To determine the change in body temperature (mean δ Temp ⁰C) at which shivering occur | 1 year
  To assess average temperature drop in order for shivering to occur from linear graph
To determine if higher OT temperature range with IV Ondansetron (HO group) is superior to individual intervention alone in reducing the incidence of PSS | 1 year
  Assessment of patient's shivering grade according to Crossley and Mahajan classification

CONTACTS AND LOCATIONS:
Overall Officials: SIU MIN LIM, L, Principal Investigator — MALAYA UNIVERSITY; SOOK HUI CHAW, AP, Study Director — MALAYA UNIVERSITY; CAROLYN YIM CHUE WAI, AP, Study Director — MALAYA UNIVERSITY; JAUHARATUNNUR ISHAK, M, Study Chair — MALAYA UNIVERSITY; TSYR XIANG TEOH, M, Study Chair — MALAYA UNIVERSITY
Locations (1):
- University Malaya Medical Center, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
All volunteers identity will be kept anonymous. However demographic data, body biometrics, underlying co-morbidities, indications for cesarean section, and study outcomes will be analysed and tabulated for publication purposes.

REFERENCES:
- [Result] Crowley LJ, Buggy DJ. Shivering and neuraxial anesthesia. Reg Anesth Pain Med. 2008 May-Jun;33(3):241-52. doi: 10.1016/j.rapm.2007.11.006. PMID 18433676
- [Result] Choi KE, Park B, Moheet AM, Rosen A, Lahiri S, Rosengart A. Systematic Quality Assessment of Published Antishivering Protocols. Anesth Analg. 2017 May;124(5):1539-1546. doi: 10.1213/ANE.0000000000001571. PMID 27622717
- [Result] Horn EP, Schroeder F, Gottschalk A, Sessler DI, Hiltmeyer N, Standl T, Schulte am Esch J. Active warming during cesarean delivery. Anesth Analg. 2002 Feb;94(2):409-14, table of contents. doi: 10.1097/00000539-200202000-00034. PMID 11812709
- [Result] Alfonsi P. Postanaesthetic shivering. Epidemiology, pathophysiology and approaches to prevention and management. Minerva Anestesiol. 2003 May;69(5):438-42. PMID 12768180
- [Result] Varshney RK, Garg M, Kapoor K, Jheetay GS. The role of ramosetron in the prevention of post-spinal shivering in obstetric patients. A prospective randomized double blind study. Rom J Anaesth Intensive Care. 2019 Apr;26(1):37-43. doi: 10.2478/rjaic-2019-0006. PMID 31111094